CLINICAL TRIAL: NCT07113353
Title: Non-Invasive Intracranial Pressure Waveform Dynamics
Brief Title: Non-Invasive ICP Monitoring Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Noah Jouett, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU20251318
Record Dates: First submitted 2025-07-29; First posted 2025-08-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Brain4Care — Non-invasive intracranial pressure monitor

SUMMARY:
Measuring the pressure inside the skull, which is called intracranial pressure, is important to treat severe neurological illness. Currently, measuring intracranial pressure requires doctors to place an invasive pressure monitor. Recently, a non-invasive intracranial pressure monitor has been developed. This monitor has a tiny pin that is placed on the head which measures the tiny movements of the skull every time the heart beats. This produces a waveform that looks very similar to an invasive intracranial pressure waveform. However, we don't know enough about how the non-invasive device to make it clinically useful yet.

DETAILED DESCRIPTION:
Assessment of intracranial pressure (ICP) is essential in the practice of neurocritical and neurosurgical care. ICP is best assessed through direct measurement with an invasive monitor, usually done by drilling a burr hole in the skull and inserting a monitor into the brain parenchyma or a catheter into the lateral ventricle. In the absence of an invasive ICP monitor, clinicians must currently rely solely on signs and symptoms of elevated ICP (e.g. alterations in pupillary constriction to light, reduced sensorium, nausea/vomiting, etc.), which occur late in the evolution of an ICP crisis. An FDA-cleared (FDA number K240821) non-invasive ICP monitor (nICPm) has been developed by Brain4Care (Johns Creek, GA). The device is equipped with piezoelectric sensors that can detect the tiny pulsations in skull expansion with every heartbeat which corresponds to the ICP waveform. Although the nICPm does not measure ICP per se, the waveform it detects is equivalent to an ICP waveform derived from an invasive monitor and has been validated to reflect intracranial pressure. Analysis of the nICPm waveform consists of factors including the P2/P1 ratio, which is the ratio of the percussive peak and the reflective peak of the ICP waveform, and time to peak (TTP), which is the time it takes for the ICP to reach maximum amplitude. nICPm waveform analysis has been studied in various clinical contexts-but how the waveform changes in response to various ICP-lowering maneuvers is incompletely characterized. Hence the current study will investigate how the nICPm waveform behaves in patients undergoing various ICP lowering procedures as a part of their ordinary, standard-of-care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18) undergoing craniotomy for any indication requiring hyperosmolar agents as a part of their surgery
* Adult patients (age >18) in the neuro-oncology or neurosurgery clinic who are receiving diagnostic/therapeutic lumbar puncture as a part of their ordinary care
* Adult patients (age >18) in the neurosurgery clinic with ventriculo-peritoneal shunts who require adjustments to increase or decrease drainage of cerebrospinal fluid.

Exclusion Criteria:

* Age <18
* Lacking capacity to provide informed consent on their own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
P2/P1 Ratio | Subject enrollment to study completion up to 100 weeks

IPD SHARING:
Plan to Share IPD: No